CLINICAL TRIAL: NCT00001960
Title: Controlled Cross-Over Study of DDD Pacemaker Therapy in Symptomatic Children With Obstructive Hypertrophic Cardiomyopathy
Brief Title: Studying the Effectiveness of Pacemaker Therapy in Children Who Have Thickened Heart Muscle
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 000007; 00-H-0007
Record Dates: First submitted 2000-01-18; First posted 2000-01-19 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2002-12

CONDITIONS: Hypertrophic Cardiomyopathy
Keywords: HCM; Pediatric; Pacemaker; Treatment; Symptoms
MeSH Terms: conditions — Cardiomyopathy, Hypertrophic

INTERVENTIONS:
Device: Pacemaker therapy

SUMMARY:
A heart condition called hypertrophic cardiomyopathy (HCM) causes abnormal thickening of the heart muscle, which obstructs the flow of blood out of the heart. The thickened muscle and the obstruction of blood flow are believed to cause chest discomfort, breathlessness, fainting, and a sensation of heart pounding. Treatment options for children with HCM include medicine, heart operation, and cardiac transplantation. However, there is no evidence that medicine prevents further thickening of heart muscle; operations carry the risk of death; and donor hearts are not always available. Several studies have shown that pacemaker treatment reduces the obstruction and improves heart complaints in patients with HCM. This study investigates further the efficacy of pacemaker treatment in children.

Patients will have exercise tests after treatment with beta blocker and verapamil and will be eligible for the study if heart complaints or reduced exercise performance continue.

A pacemaker that treats slow heart rhythms will be inserted. The patient will be sedated and local anesthesia will be administered to numb the area. The procedure takes about an hour.

The study will last two years. Patients will be placed on one of two pacemaker programs for the first year and another the second year. At 3- and 6-month follow-up visits, a pacemaker check and echocardiogram will be performed. After 1 year, patients will be admitted to NIH for 2 to 3 days for exercise tests, echocardiogram, and cardiac catheterization. Also, the pacemaker will be changed to the second program. At 15- and 18-month follow-up visits, a pacemaker check and echocardiogram will be performed. After 2 years, patients will again be admitted for 2 to 3 days for exercise tests, echocardiogram, and cardiac catheterization. A pregnancy test will be given to females of child-bearing age before each cardiac catheterization and electrophysiology study.

At the end of the study, the pacemaker will be set to the program that worked better.

Risks of pacemaker insertion include lung collapse, infection, blood vessel damage, bleeding, heart attack, and death. Risks of cardiac catheterization include infection, bleeding, blood clots, abnormal heart rhythms, perforation of the heart, need for surgery, and death. However, the safety record for both these procedures at NIH has been excellent. The radiation exposure exceeds the NIH radiation guidelines for children, but this exposure in adults has not been associated with any definite adverse effects.

DETAILED DESCRIPTION:
Studies suggest that DDD pacemaker therapy is effective in improving symptoms and reducing intra-ventricular pressures and pressure gradients in children with obstructive HCM during a period of rapid body growth when the severity of the disease is expected to worsen. We propose a randomized, cross-over study of DDD pacing versus placebo (AAI pacing mode) in children who have limited exercise performance and/or symptoms despite medical therapy (beta-blocker or verapamil). Study subjects will receive a pacemaker and will be randomized to one of two pacing modes (DDD, AAI). After a 1-year follow-up evaluation the children will cross-over to the alternative pacing mode, and will be re-evaluated after a further year. All children will continue to receive optimum medical therapy (beta-blocker or verapamil) based on improvement in symptoms and exercise performance. The subjects will undergo outpatient evaluations (exercise tests and echocardiography) 3, 6, 15, and 18 months after pacemaker implantation, and inpatient evaluations (exercise tests, echocardiography, and cardiac catheterization) 1 year and 2 years after entry into the study. Primary end-points will be exercise duration and severity of LV outflow obstruction. The patient, parents, referring physician, and individual supervising the exercise tests will be blinded to the pacing mode.

ELIGIBILITY:
INCLUSION CRITERIA:

Children of either gender, aged 4 to 18 years.

Obstructive HCM defined as LV hypertrophy, and an LV intra-cavitary pressure gradient measured at cardiac catheterization of greater than or equal to 30 mm Hg at rest or greater than or equal to 50 mm Hg following isoproterenol infusion to a heart rate of greater than or equal to 100 beats per minute.

Cardiac symptoms (chest discomfort, dyspnea, lightheadedness or presyncope, syncope, cardio-respiratory arrest, palpitations, excessive fatigue); and/or exercise duration which is less than 10th percentile predicted for age/gender despite a trial of a beta-blocker therapy and a trial of verapamil therapy.

EXCLUSION CRITERIA:

Other systemic diseases that prevent assessment by exercise tests and cardiac catheterization.

Chronic atrial fibrillation.

Positive pregnancy test: A negative urine pregnancy test will be required before each cardiac catheterization, electrophysiologic study and thallium study. Pregnant or lactating subjects may not participate in the study due to potential teratogenic effects of radiation.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50
Dates: Start 1999-11; Study Completion 2002-12

CONTACTS AND LOCATIONS:
Locations (1):
- National Heart, Lung and Blood Institute (NHLBI), Bethesda, Maryland, United States

REFERENCES:
- [Background] Fananapazir L, Chang AC, Epstein SE, McAreavey D. Prognostic determinants in hypertrophic cardiomyopathy. Prospective evaluation of a therapeutic strategy based on clinical, Holter, hemodynamic, and electrophysiological findings. Circulation. 1992 Sep;86(3):730-40. doi: 10.1161/01.cir.86.3.730. PMID 1516184
- [Background] Wigle ED, Rakowski H, Kimball BP, Williams WG. Hypertrophic cardiomyopathy. Clinical spectrum and treatment. Circulation. 1995 Oct 1;92(7):1680-92. doi: 10.1161/01.cir.92.7.1680. PMID 7671349
- [Background] Fananapazir L. Advances in molecular genetics and management of hypertrophic cardiomyopathy. JAMA. 1999 May 12;281(18):1746-52. doi: 10.1001/jama.281.18.1746. No abstract available. PMID 10328076